CLINICAL TRIAL: NCT01168583
Title: Investigation of the Effect of Post-operative Fluid Balance on Inflammatory Mediators in Patients Undergoing Cardiovascular Surgery
Brief Title: Fluid Balance and Clinical Outcomes
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 126-2010
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Fluid Balance; Input and Output; Inflammatory Mediators; Acute Kidney Injury; Mortality
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive Fluid Balance of 2000ml
- Negative Fluid Balance of 2000ml

SUMMARY:
This study is about investigating the relationship of postoperative fluid balance, inflammation and acute kidney injury. This is a non-interventional study (no drug administration). The investigators will collect baseline demographic data, postoperative fluid balance status by Intake-output data, follow routine labs and collect 1 blood sample (0.5ml) with morning lab draws on day 1 and 5ml urine samples on day 1 and 2.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older, and
* Undergoing elective cardiothoracic surgery(s), alone or in combination with other procedures/surgery(s): thoracic aortic aneurysm, cardiac valves, coronary artery bypass grafting, abdominal thoracic aneurysm, and other cardiovascular surgery.

Exclusion Criteria:

* Pregnancy
* History of any organ transplant
* Preoperative intra-aortic balloon pump (IABP)
* Current use of natriuretic peptides
* ESRD patients on dialysis
* Estimated GFR < 30ml/min using MDRD equation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the hospital for elective cardiothoracic surgery.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2010-07; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: A Ahsan Ejaz, M.D, Principal Investigator — University of Florida; Ganesh Kambhampati, M.D, Principal Investigator — University of Florida
Locations (1):
- Shands Hospital, University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Kambhampati G, Ejaz NI, Asmar A, Aiyer RK, Arif AA, Pourafshar N, Yalamanchili VR, Ejaz AA. Fluid balance and conventional and novel biomarkers of acute kidney injury in cardiovascular surgery. J Cardiovasc Surg (Torino). 2013 Oct;54(5):639-46. PMID 24002394
- [Derived] Ejaz AA, Kambhampati G, Ejaz NI, Dass B, Lapsia V, Arif AA, Asmar A, Shimada M, Alsabbagh MM, Aiyer R, Johnson RJ. Post-operative serum uric acid and acute kidney injury. J Nephrol. 2012 Jul-Aug;25(4):497-505. doi: 10.5301/jn.5000173. PMID 22684655
- [Derived] Kambhampati G, Ross EA, Alsabbagh MM, Asmar A, Pakkivenkata U, Ejaz NI, Arif AA, Ejaz AA. Perioperative fluid balance and acute kidney injury. Clin Exp Nephrol. 2012 Oct;16(5):730-8. doi: 10.1007/s10157-012-0623-5. Epub 2012 Mar 29. PMID 22457087